CLINICAL TRIAL: NCT03829020
Title: An Open-Label Phase 1 Study of Metformin and Nelfinavir in Combination With Bortezomib in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Metformin, Nelfinavir, and Bortezomib in Treating Patients With Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1811; NCI-2019-00466 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1811 (Other: Mayo Clinic in Rochester); 18-000858 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Metformin; Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (metformin, nelfinavir) (Experimental): Patients receive metformin hydrochloride PO on days 1-14, nelfinavir mesylate PO BID on days 1-14, and bortezomib SC on days 1, 8, and 15. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Metformin Hydrochloride; Drug: Nelfinavir Mesylate

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Metformin Hydrochloride — Given PO
  Other Names: APO-Metformin; Cidophage; Dimefor; Glifage; Glucoformin; Glucophage; Glucophage ER; Metformin HCl; Riomet; Siofor
Drug: Nelfinavir Mesylate — Given PO
  Other Names: AG1343; Viracept

SUMMARY:
This phase I trial studies the side effects and best dose of metformin and nelfinavir in combination with bortezomib in treating patients with multiple myeloma that has come back or does not respond to treatment. Metformin may stop the growth of tumor cells by disrupting the energy source within multiple myeloma cells. Nelfinavir and bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving metformin, nelfinavir, and bortezomib may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the maximum tolerated dose (MTD) of administering metformin hydrochloride (metformin) and nelfinavir mesylate (nelfinavir) in combination with bortezomib in patients with relapsed/refractory multiple myeloma.

SECONDARY OBJECTIVES:

I. To describe the safety and tolerability of metformin and nelfinavir in combination with bortezomib in patients with relapsed/refractory multiple myeloma.

II. To assess the best hematological response of the combination of metformin, nelfinavir and bortezomib within 6 cycles of initiating therapy.

EXPLORATORY OBJECTIVE:

I. Assess clinical biomarkers predictive of response to the combination of metformin, nelfinavir and bortezomib such as bioenergetic profiles of the myeloma cells, GLUT4 expression on myeloma cells, PI3K/AKT/mTOR and MAPK signaling pathways and metabolomics-based profiling.

OUTLINE: This is a dose-escalation study of metformin hydrochloride and nelfinavir mesylate.

Patients receive metformin hydrochloride orally (PO) on days 1-14, nelfinavir mesylate PO twice daily (BID) on days 1-14, and bortezomib subcutaneously (SC) on days 1, 8, and 15. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Actively relapsing multiple myeloma
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 0.5 g/dL

    * If immunoglobulin A (IgA) isotype, then IgA quantification > upper limit of normal
  * >= 200 mg of monoclonal protein in the urine on 24-hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis >= 10% (evaluable disease)
* Patients must have received at least 2 prior regimens and patients should have been exposed to a proteasome inhibitor (PI), an immunomodulatory drugs (IMiD) and an anti-CD38 antibody. NOTE: Induction therapy followed by an autologous stem cell transplant (ASCT) and maintenance therapy without any relapse counts as 1 regimen
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Hemoglobin >= 8.0 g/dL (No red cell transfusion should have been administered within 4 days of registration) (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 50,000/mm^3 or >= 30,000/mm^3 if bone marrow plasma cells percentage >= 50% by morphology (No platelet transfusion should have been administered within 7 days of registration) (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =< 14 days prior to registration)
* Calculated creatinine clearance >= 45 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only. NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Provide written informed consent
* Able to swallow metformin and nelfinavir tablets
* Willingness to provide mandatory blood sample and bone marrow aspirate for research purposes
* Willingness to return to Mayo Clinic for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* The following populations should be excluded from study:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Major surgery =< 14 days before study registration
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Another active malignancy requiring therapy such as radiation, chemotherapy, or immunotherapy. NOTE: Patients on hormonal therapy for treated breast or prostate cancer are permitted if they meet other eligibility criteria
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Known allergy to any of the study medications, their analogues or excipients in the various formulations
* Subjects must not have conditions associated with increased risk of metformin associated lactic acidosis, including New York Heart Association class III or IV congestive heart failure, history of acidosis of any type, alcoholic liver disease, or habitual intake of 3 or more alcoholic beverages per day
* Clinical history of type I or type II diabetes
* Currently on either metformin or a HIV-PI or both
* Elevated baseline lactate level > ULN (2.3 mmol/L)
* Any of the following recent prior anti-myeloma therapy:

  * Alkylators (e.g. melphalan, cyclophosphamide) and anthracyclines =< 14 days prior to registration
  * High dose corticosteroids (equivalent to > 10 mg of prednisone/day) and immunomodulatory drugs (thalidomide or lenalidomide) =< 7 days prior to registration
  * Monoclonal antibodies =< 14 days prior to registration
* Currently receiving sensitive/moderate sensitive substrates of CYP3A4, strong CYP3A4 inhibitors, or strong CYP3A4 inducers that cannot be discontinued 7 days prior to starting study and throughout study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of the combination of metformin, nelfinavir, and bortezomib | 42 days
  Defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients (at least 2 of a maximum of 6 new patients).

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2.5 years
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Hematologic response rate | Up to 2.5 years
  Defined to be a stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) noted as the objective status on two consecutive evaluations. Exact binomial 95% confidence intervals for the true hematologic response rate will be calculated.

OTHER OUTCOMES:
Clinical biomarker analysis | Up to 2.5 years
  Will be explored and correlated with response to the combination of metformin, nelfinavir, and bortezomib using Fisher's exact and Wilcoxon rank sum tests. Clinical biomarkers examined may include bioenergetic profiles of the myeloma cells, GLUT4 expression on myeloma cells, PI3K/AKT/mTOR and MAPK signaling pathways and metabolomics-based profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson I. Gonsalves, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials